CLINICAL TRIAL: NCT00810706
Title: A Phase III Randomized Parallel-Group Multicenter Trial, Designed to Compare 5 Years of Adjuvant Exemestane Versus 5 Years of Observation in Postmenopausal Women With Operable Breast Cancer Who Have Received 5-7 Years of Adjuvant Tamoxifen.
Brief Title: Adjuvant Post-Tamoxifen Exemestane Trial
Acronym: ATENA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Publication of MA17 results (similar trial in the extented adjuvant setting with letrozole)
Sponsor: Hellenic Breast Surgeons Society (Other)
Responsible Party: Markopoulos Christos, Hellenic Breast Surgeons Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 971-ONC-0028-085
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Aromatase inhibitors; Exemestane; Tamoxifen; Lipids
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: observation only (No Intervention): Patients have completed at least 5 years and not more than 7 years of continued treatment with tamoxifen (20 mg/day). Tamoxifen could have been discontinued up to 6 months prior to study entry.
- 2: Exemestane (Active Comparator): Patients randomised to receive exemestane (25 mg/day) for 5 years, following completion of 5-7 years of Tamoxifen treatment
  Interventions: Drug: exemestane

INTERVENTIONS:
Drug: exemestane — Patients randomised to receive exemestane (25 mg/day) for 5 years.
  Other Names: Aromasin
  Arms: 2: Exemestane

SUMMARY:
The ATENA phase III randomized parallel-group multicenter trial is designed to compare 5 years of adjuvant exemestane versus 5 years of observation in postmenopausal women with operable breast cancer who have received 5-7 years of adjuvant tamoxifen. The primary endpoint for the core protocol is disease-free survival (DFS). Exemestane treatment is planned for 5 years unless disease relapse or excessive toxicity is documented, the patient refuses further treatment or any new anti-cancer therapy is initiated.

DETAILED DESCRIPTION:
* Patients must have completed at least 5 years and not more than 7 years of continued treatment with tamoxifen (20 mg/day), while tamoxifen could have been discontinued up to 6 months prior to study entry.
* A substudy (ATENA lipid substudy)is designed to evaluate changes in the patients' serum lipid profile during study treatment.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women only
* histologically confirmed stage I-IIIA primary adenocarcinoma of the breast
* estrogen and/or progesterone receptors positive or unknown
* patients should have undergone surgery with a curative intent
* patients must have completed at least 5 years and not more than 7 years of continued treatment with tamoxifen (20 mg/day), while tamoxifen could have been discontinued up to 6 months prior to study entry
* Absence of any evidence of local or distant metastatic disease was required prior to randomization

Exclusion Criteria:

* DCIS, bilateral breast cancer, evidence of metastasis, ER and Pgr negative

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2001-04; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
DFS | 5 years

SECONDARY OUTCOMES:
effect of exemestane on lipaemic profile | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Breast Surgeons Society, Athens, Greece

REFERENCES:
- [Result] Markopoulos C, Chrissochou M, Michailidou A, Tzoracoleftherakis E, Xepapadakis G, Papadiamantis J, Misitzis J, Zobolas V, Bafaloukos D, Gogas H. Effect of exemestane on the lipidemic profile of post-menopausal operable breast cancer patients following 5-7 years of adjuvant tamoxifen: preliminary results of the ATENA substudy. Anticancer Drugs. 2005 Sep;16(8):879-83. doi: 10.1097/01.cad.0000173478.12981.e1. PMID 16096437
- [Result] Markopoulos C, Chrissochou M, Antonopoulou Z, Xepapadakis G, Papadiamantis J, Tzoracoleftherakis E, Gogas H. Duration of tamoxifen effect on lipidemic profile of postmenopausal breast cancer patients following deprivation of treatment. Oncology. 2006;70(4):301-5. doi: 10.1159/000096251. Epub 2006 Oct 12. PMID 17047401
- [Derived] Markopoulos C, Dafni U, Misitzis J, Zobolas V, Tzoracoleftherakis E, Koukouras D, Xepapadakis G, Papadiamantis J, Venizelos B, Antonopoulou Z, Gogas H. Extended adjuvant hormonal therapy with exemestane has no detrimental effect on the lipid profile of postmenopausal breast cancer patients: final results of the ATENA lipid substudy. Breast Cancer Res. 2009;11(3):R35. doi: 10.1186/bcr2320. Epub 2009 Jun 16. PMID 19531217